CLINICAL TRIAL: NCT07162753
Title: Detection of Racial Bias in an Artificial Intelligence Based Orthodontic Diagnosis System
Brief Title: Assesment of Ethnic Bias in an Artificial Intelligence Based Orthodontic Diagnosis System
Status: Recruiting | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Collaborators: PEBS DENTAL CLINIC (Unknown)
Responsible Party: Principal Investigator, Aslı Eker Davut, Dentist - PhD Student, Bezmialem Vakif University
Other Study IDs: E-54022451-050.04-177270
Record Dates: First submitted 2025-08-26; First posted 2025-09-09 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-07

CONDITIONS: Class I Malocclusion; Class II Div 1 Malocclusion; Class II Division 2 Malocclusion; Class III Malocclusion
Keywords: Artificial Intelligence; Deep Learning; Ethnic Bias; Machine Learning; Orthodontics
MeSH Terms: conditions — Malocclusion, Angle Class I; Malocclusion, Angle Class II; Malocclusion, Angle Class III

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Turkish Citizen's Control Group (Hold-out): The AI system was trained with data from 7,000 people. To test whether the AI has bias, the system should be evaluated both on a group of Turkish citizens who were not included in the training data and on patients from different ethnic backgrounds.
- Individuals from different ethnic backgrounds: Test set, consisting of individuals from different ethnic backgrounds.

SUMMARY:
This study explores how artificial intelligence (AI) can be used in orthodontics, which is the area of dentistry that focuses on correcting jaw and bite problems. AI is a computer technology that can learn from large amounts of data and then make predictions or decisions. It is already being tested in medicine and dentistry to help doctors and dentists diagnose conditions.

For this study, the AI system was trained using photographs and X-rays from patients in Turkey. The system learned to recognize specific orthodontic skeletal malocclusions. After the training stage, the AI was tested in two groups: one group included Turkish patients whose records were not used in training, and the other group included patients from different ethnic backgrounds who were treated at a clinic in Belgium. This design allows researchers to see if the AI works equally well for people of different backgrounds.

Only photographs and X-rays taken before orthodontic treatment are used in the study, and all data are anonymized so that no personal information is shared. The images must meet certain quality standards. For example the head must be in natural position, with no beards, scars, or previous orthodontic treatment that might affect the image. Patients who do not meet these criteria are not included.

The AI program analyzes the profile photographs, prepares them for evaluation by adjusting and standardizing the images, and then tries to decide each patient has which malocclusion. The results from Turkish patients and patients from other ethnic groups are compared to see if the system makes fair and accurate decisions for everyone.

The purpose of this study is not to test a new treatment, but to understand how well AI can recognize orthodontic problems in different populations. This information is important because AI systems are increasingly being used in healthcare, and they need to be fair and accurate for all patients, not just those from one group.

By participating, patients help researchers learn whether AI in orthodontics is reliable across diverse communities. This knowledge can guide future improvements in AI technology, ensuring that it supports orthodontists in providing safe, equal, and effective care for everyone.

DETAILED DESCRIPTION:
This study investigates how artificial intelligence (AI) can be used to diagnose skeletal malocclusions. AI is a computer technology that can learn from data, recognize patterns, and then make predictions. It is already being used in different areas of medicine and dentistry, but its accuracy and fairness may depend on the data it was trained with.

In orthodontics, skeletal problems are usually classified into four main groups: Class I (normal skeletal relationship), Class II Division 1, Class II Division 2 (upper jaw forward or lower jaw retruded or both ), and Class III (lower jaw forward in relation to the upper jaw or upper jaw retruded relation to lower jaw or both).

For this study, an AI system was trained with profile photographs and X-rays of 3,280 Turkish patients. The system learned to recognize all four types of skeletal relationships: Class I, Class II Division 1, Class II Division 2, and Class III. After the training, the AI was tested on new groups of patients whose images were not part of the training set. This included a group of Turkish patients and another group of patients from different ethnic backgrounds treated in Belgium. By comparing the AI's results in these two groups, researchers will be able to see whether the system works equally well for people of different ethnicities.

The patient data used in this study is completely anonymized. Only pre-treatment profile photographs and lateral cephalometric X-rays are included. The images must comply with quality standards such as being taken in natural head position, with a clear background and without beard, scars, or previous orthodontic treatment that might interfere with recognition. Patients whose photographs do not meet these standards are excluded.

This research is conducted as a cross-sectional diagnostic accuracy study (single-gate, multi-center). The diagnostic performance of the AI system is evaluated using accuracy, recall (sensitivity), precision, false positive rate, F1 score, and area under the curve (AUC).

The aim of this study is to evaluate whether an AI-based system used by patients for orthodontic diagnosis provides fair and reliable results across different ethnic groups.

ELIGIBILITY:
* Patients with lateral profile photographs taken before starting orthodontic treatment
* Profile photographs with a plain background
* Patient in natural head position facing forward
* No beard or mustache that could camouflage the profile
* Availability of lateral cephalometric radiographs taken before treatment together with the profile photograph

Exclusion criteria:

* Blurry missing or non standard profile photographs
* Presence of beard mustache scars cleft lip palate or soft tissue deformities that may significantly affect facial appearance
* Previous orthodontic treatment history

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: One group consists of Turkish citizens who were not included in the AI training set. Another group consists of patients who visited the PEBS clinic in Brussels, Belgium, representing individuals from different ethnic backgrounds.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-08-11 (Estimated)

PRIMARY OUTCOMES:
Accuracy | At baseline (retrospective single time-point data analysis)
  Accuracy (proportion of correctly classified cases) will be compared between Turkish test set, and non-Turkish cohort from different ethnic backgrounds.

SECONDARY OUTCOMES:
Precision (Positive Predictive Value) | At baseline (retrospective single time-point data analysis)
  Percentage of cases labeled as Class III by AI that are truly Class III. Rate of AI-predicted positive cases that are truly positive, compared between Turkish group and non-Turkish ethnic group
Recall | At baseline (retrospective single time-point data analysis)
  Percentage of true Class III cases correctly identified by AI
False Positive Rate | At baseline (retrospective single time-point data analysis)
  Rate of negative cases incorrectly classified as positive by AI, compared across cohorts.
F1 score | At baseline (retrospective single time-point data analysis)
  Harmonic mean of precision and recall (range 0-1). Higher values indicate better overall performance, while lower values indicate poor balance between sensitivity and precision.

CONTACTS AND LOCATIONS:
Overall Officials: Banu Kılıç, Doctor of Orthodontics, Study Director — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakıf University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared on reasonable request to the corresponding author.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 3 months and ending a year after the publication of results
Access Criteria: The investigators can access to the corresponding author by e-mail.

REFERENCES:
- [Background] Allareddy V, Oubaidin M, Rampa S, Venugopalan SR, Elnagar MH, Yadav S, Lee MK. Call for algorithmic fairness to mitigate amplification of racial biases in artificial intelligence models used in orthodontics and craniofacial health. Orthod Craniofac Res. 2023 Dec;26 Suppl 1:124-130. doi: 10.1111/ocr.12721. Epub 2023 Oct 17. PMID 37846615
- [Background] Kilic B, Ibrahim AH, Aksoy S, Sakman MC, Demircan GS, Onal-Suzek T. A family-centered orthodontic screening approach using a machine learning-based mobile application. J Dent Sci. 2024 Jan;19(1):186-195. doi: 10.1016/j.jds.2023.05.001. Epub 2023 May 17. PMID 38303845